CLINICAL TRIAL: NCT01778920
Title: Intraoperative Imaging of Pulmonary Adenocarcinoma
Brief Title: Pilot and Feasibility Study of the Imaging Potential of EC17: Intraoperative Folate-fluorescein Conjugate (EC17) Lung Cancer (CA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 815058; EC17 Lung Cancer (Other: University of Pennsylvania)
Record Dates: First submitted 2013-01-18; First posted 2013-01-29 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2015-12

CONDITIONS: Lung and Pleural Malignancies; Neoplasms; Nodules; Adenocarcinoma
MeSH Terms: conditions — Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV Injection of EC17 (Experimental): The group will receive a single dose of EC17, infused over 10 minutes, prior to surgery. Then, during surgery, the EC-17 will be imaged with a camera that the investigators have developed.
  Interventions: Drug: EC17 imaging contrast agent

INTERVENTIONS:
Drug: EC17 imaging contrast agent — This is an imaging agent to locate lung adenocarcinoma cancer cells during surgery

SUMMARY:
The goal of this study is to perform imaging of patient's tumors while the chest is open and the tumor is being removed.

According to the World Health Organization, lung cancer is the most common cause of cancer-related death in men and women, and is responsible for 1.3 million deaths worldwide annually as of 2004. Surgery remains the best option for patients presenting with operable Stage I or II cancers, however the five year survival rate for these candidates remains at a dismal 53% for Stage I and 32% for Stage II. The high rates of recurrence suggest that surgeons are unable to completely detect and remove primary tumor nodules in a satisfactory manner as well as lingering metastases in sentinel lymph nodes. By ensuring a negative margin through imaging during surgery it would be possible for us to improve the rates of recurrence free patients and thus overall survival.

Thoracic malignancies are the ideal disease to investigate intra-operative imaging. Over 85% of lung and pleural malignancies express folate receptor alpha (FRA). It is important to note that FRA is expressed only in the proximal tubules of the kidneys, activated macrophages, and in the choroidal plexus. Thus, the false positive detection rate is expected to be extremely low. A group well known to us in the Netherlands has completed a pilot study utilizing a folate-fluorescein isothiocyanate (folate-FITC) conjugate in 12 patients with ovarian cancer. Another group of investigators in Mayo have subsequently performed this study on 20 more patients without any serious adverse events (personal communication). They report excellent sensitivity and specificity with this technique with only grade 1 side effects (allergic reaction). All side effects reversed when the injection was halted. Patients with a history of allergic reactions to insect bites should not participate (fluorescein is derived from the firefly insect, folate is an essential vitamin).

DETAILED DESCRIPTION:
This will identify the margins and the lymph nodes that may have cancer cells during cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Patients presenting with a lung or pleural nodule or mass presumed to be resectable on pre-operative assessment
* Good operative candidate
* Subject capable of giving informed consent and participating in the process of consent

Exclusion Criteria:

* Pregnant women as determined by urinary or serum beta human chorionic gonadotropin (hCG) within 72 hours of surgery
* Patients with a history of anaphylactic reactions to Folate-FITC or insects
* At-risk patient populations:

  * Homeless patients
  * Patients with drug or alcohol dependence
  * Children and neonates
  * Patients unable to participate in the consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of FRA tumors identified by EC17 during surgery. | Within two to four hours of injection of the EC17
  Measure the number of patients who have a positive margin during lung cancer surgery 2 - 4 hours after receiving administration of EC17.

SECONDARY OUTCOMES:
The number of participants that will have an adverse reaction to the EC17 | Day 1 - Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, Principal Investigator — Philadelphia VA Medical Center, Philadelphia, PA
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Okusanya OT, DeJesus EM, Jiang JX, Judy RP, Venegas OG, Deshpande CG, Heitjan DF, Nie S, Low PS, Singhal S. Intraoperative molecular imaging can identify lung adenocarcinomas during pulmonary resection. J Thorac Cardiovasc Surg. 2015 Jul;150(1):28-35.e1. doi: 10.1016/j.jtcvs.2015.05.014. Epub 2015 May 7. PMID 26126457